CLINICAL TRIAL: NCT04952896
Title: Using Magnetic Resonance Imaging and DL Methods to Explore the Diagnosis and Clinical Prognosis of Joint Synovitis.
Brief Title: Clinical Study of Magnetic Resonance Imaging and Deep Learning of Joint Synovial Disease
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2019168
Record Dates: First submitted 2021-06-29; First posted 2021-07-07 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-05

CONDITIONS: Synovial Diseases; Pigmented Villonodular Synovitis; Gout; Rheumatoid Arthritis
Keywords: pigmented villonodular synovitis; deep learning; knee synovitis; MRI
MeSH Terms: conditions — Synovitis, Pigmented Villonodular; Gout; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group of patients with pigmented villonodular synovitis: Diagnosis confirmed by arthroscopic pathological biopsy.
  Interventions: Diagnostic Test: Synovitis diagnosis
- Group of patients with rheumatoid arthritis: Diagnosis determined by clinical history, laboratory tests and arthroscopic pathology biopsy.
  Interventions: Diagnostic Test: Synovitis diagnosis
- Group of patients with gout: Diagnosis was determined by laboratory tests, energy spectrum imaging and arthroscopic pathology biopsy.
  Interventions: Diagnostic Test: Synovitis diagnosis

INTERVENTIONS:
Diagnostic Test: Synovitis diagnosis

SUMMARY:
Through the high-throughput feature extraction of magnetic resonance images, the deep learning prediction model of joint synovial lesions is constructed used for the diagnosis, differential diagnosis and curative effect monitoring of joint synovial lesions.

DETAILED DESCRIPTION:
The study applies magnetic resonance and deep learning (DL) to the diagnosis of joint synovial lesions, aims to have a more comprehensive understanding of the pathophysiology of the occurrence and development of joint synovial lesions. As a non-invasive imaging method to assess the condition of the disease, DL methods excavates the deep features contained in the image, quantifies the joint synovial lesions, and then gives more information to the clinician in the diagnosis and differential diagnosis of the joint synovial lesions, provide important information for the planning of individualized treatment plans for patients with joint synovial diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with joint synovial disease through radiological examination, arthroscopy or pathological biopsy of the joint, or whose clinical manifestations meet the diagnostic criteria of the American College of Rheumatology (ACR) for joint synovial disease.
2. Patients received pre-treatment MR.

Exclusion Criteria:

1. Patients who have received surgery, medication or other systemic treatment before standardized MRI scan.
2. Poor image quality.
3. Articular hemorrhage.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with joint synovial disease through radiological examination, arthroscopy or pathological biopsy of the joint, or whose clinical manifestations meet the diagnostic criteria of the American College of Rheumatology (ACR) for joint synovial disease.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Patient's diagnosis | 2019-2022
  Type of synovitis disease in patients with a clear comprehensive diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University third hospital, Beijing, Please Select An Option Below, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, Analytic Code